CLINICAL TRIAL: NCT04297475
Title: The Clinical Feasibility and Added Value of a Multi-modal Photoacoustic/Ultrasonic Imaging System in the Evaluation of Rheumatoid Arthritis
Brief Title: The Clinical Feasibilityof a Multi-modal Photoacoustic/Ultrasonic Imaging System in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: MMPAUS RA
Record Dates: First submitted 2019-07-13; First posted 2020-03-05 (Actual); Last update posted 2020-10-28 (Actual); Status verified 2020-09

CONDITIONS: Rheumatoid Arthritis; Ultrasonography
Keywords: rheumatoid arthritis; ultrasonography; multi-modal imaging; photoacoustic imaging
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- rheumatoid arthritis: The patients are diagnosed with RA according to the American College of Rheumatology (ACR) criteria, and the current clinical state was in-active or relapse. The patients receive final diagnosis and disease evaluation by two experienced rheumatologists
  Interventions: Diagnostic Test: Multi-modal photoacoustic/ultrasonic (PA/US) imaging system

INTERVENTIONS:
Diagnostic Test: Multi-modal photoacoustic/ultrasonic (PA/US) imaging system — The multi-modal PA/US imaging system is equipped with a handheld 3D PA/US probe, and able to provide 3D volume data of dual-wavelength PA imaging of small joints, in addition to real-time 2D PA/US imaging.

SUMMARY:
New type of imaging method is in demand clinically for early detection and treatment guiding of RA. Photoacoustic imaging (PAI), a hot spot in medical imaging society, which combines the merits of optical imaging and US and has a capacity in morphological, functional and molecular imaging, has shown potential in visualizing superficial organs, including small joints. The investigators developed a multi-modal photoacoustic/ultrasound (PA/US) imaging system, equipped with a handheld 3D PA/US probe, which wass able to provide 3D volume data of dual-wavelength PA imaging of small joints, in addition to real-time 2D PA/US imaging. The investigators plan to recruit RA patients in different disease conditions and healthy volunteers to receive the 2D and 3D PA/US examination on the 2nd and 3rd MCP, PIP joints and wrist joints using this imaging system, and to evaluate the potential clinical role of the imaging system in RA, and its added value to current imaging methods.

DETAILED DESCRIPTION:
The multi-modal PA/US imaging system was built on a high-end commercial US platform, and allowed real-time imaging of grey-scale US imaging, Color-Doppler US (CDUS) imaging and dual-wavelength PA imaging. The PA/US images were acquired using a hand-held probe integrated optical devices and US transducers. 3D volume data of the selected joint of each participant was collected using an automatic scanning device after the dual-modal imaging. The investigators plan to recruit RA patients from the outpatient department of Rheumatology of our hospital, who have been diagnosed as RA by experienced rheumatologists. The patients and healthy volunteers will receive multi-modal imaging examinations using the novel imaging system. The MCP 2 and 3, PIP 2 and 3, and wrist of bilateral hand were chosen for the multi-modal imaging. Conventional US scanning of the joints, including grey-scale US, CDUS, and PDUS, will be carried out by an experienced US operator. Afterwards, 2D and 3D PA/US imaging will be implemented for each joint by the same operator. All of the imaging data will be analysed by the Matlab software.

ELIGIBILITY:
The inclusion criteria

1. The patients were above 18 years-old;
2. The patients were diagnosed with RA according to the American College of Rheumatology (ACR) criteria, and the current clinical state was in-active or relapse;
3. The patients were consent to receive examinations of photoacoustic imaging.

The exclusion criteria

1. The patients had mental disease or other severe diseases, and were not capable of receiving imaging examinations;
2. The patients had strong reaction to laser light.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The RA patients are diagnosed as RA by two experienced rheumatologists.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
The PA scores of 50 participants with RA identified by the multi-modal imaging system are in accordance with clinical scoring | 3-6 months
  A total of 50 participants received semi-quantitatively measurement of PA signals by the imaging system using a 0-3 scoring system. Score 0 is no PA signals, which represents no detectable active inflammation on PA imaging. Score 1 means less than 3 bars of PA signals within the inflamed regions. Score 2 means multiple PA signals within less than half of the inflammatory lesions. And score 3 means abundant PA signals in over half of the lesions of RA synovium or tenosynovium, which may represent high inflammation activity.
The functional imaging of 60 RA patients assessed by the multi-modal imaging system | 12-15 months
  The oxgenation levels of local joint tissues of 60 RA patients are measured by dual-wavelength PA imaging.

CONTACTS AND LOCATIONS:
Overall Officials: Yuxin Jiang, Doctor, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Yang M, Zhao C, Wang M, Wang Q, Zhang R, Bai W, Liu J, Zhang S, Xu D, Liu S, Li X, Qi Z, Yang F, Zhu L, He X, Tian X, Zeng X, Li J, Jiang Y. Synovial Oxygenation at Photoacoustic Imaging to Assess Rheumatoid Arthritis Disease Activity. Radiology. 2023 Jan;306(1):220-228. doi: 10.1148/radiol.212257. Epub 2022 Aug 23. PMID 35997608